CLINICAL TRIAL: NCT07237516
Title: Zymfentra (Infliximab-dyyb) REal World Cohort STudy
Acronym: ZEST
Status: Recruiting | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Celltrion (Industry)
Responsible Party: Sponsor
Other Study IDs: 25-2184
Record Dates: First submitted 2025-11-03; First posted 2025-11-19 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Ulcerative Colitis (UC); Crohn's Disease (CD); Indeterminate Colitis; Inflammatory Bowel Disease (IBD)
Keywords: Zymfentra; ZEST
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease; Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to learn about how effective Zymfentra (IFX=dyyb) is when treating patients with Crohn's disease (CD) and ulcerative colitis (UC) Does Zymfentra lead to a reduction in symptoms at intervals throughout one year? Participants being prescribed Zymfentra (IFX-dyyb as part of their regular medical care for CD or UC will answer online survey questions about their bowel habits for 1 year.

ELIGIBILITY:
Inclusion Criteria:

- 1. Adult patients, age 18 years or older, with Crohn's disease (CD), ulcerative colitis (UC) or Inflammatory Bowel Disease Unclassified (IBDU), who are either starting Zymfentra at week 10 (IFX-dyyb) in the setting of standard-of-care initiation with intravenous Infliximab (IFX) originator or IFX biosimilars induction therapy at weeks 0,2,6 or switching from intravenous IFX originator or IFX biosimilars during maintenance therapy to Zymfentra (IFX-dyyb) 2. Anticipation that the patient will be followed by the participating center for the next 12 months.

3. Diagnosis of CD, UC or IBDU must be established based on standard clinical, radiographic, endoscopic, and histologic criteria as described below.

The following diagnostic criteria were developed by the NIDDK IBD Genetics Consortium and are provided as guidelines to complete documentation on individuals with CD, UC or IBDU:

A) Symptoms including one or more: diarrhea, rectal bleeding, abdominal pain, fever, complicated perianal disease, extraintestinal manifestations, weight loss or failure to thrive.

AND B) Symptoms on two or more occasions separated by at least 8 weeks or ongoing symptoms of at least 6 weeks duration. When there has been a single episode of colitis (in some instances less than 6 weeks duration) resulting in colectomy and resolution of disease symptoms, pathology on the colectomy specimen should be consistent with idiopathic IBD and microbiology studies should be negative.

AND

C) One or more of the following providing objective evidence of inflammation:

Endoscopic: Mucosal edema, erythema, loss of normal submucosal vasculature, friability, ulceration, stricture formation, pseudopolyps, mucosal edema, erythema. Where there are only minor changes (mucosal edema, erythema, loss of normal submucosal vasculature, friability) mucosal biopsies should have been done to confirm the presence of IBD.

Radiologic: Mucosal thickening and/or nodularity, ulceration, stricture, pseudopolyps, fistula formation, pseudosacculation. Minor changes alone (mucosal thickening and/or nodularity) should not be sufficient to make a diagnosis of IBD.

Histologic: Mucosal erosion or ulceration, architectural changes of crypts, Paneth cell metaplasia (in colon), transmural inflammatory infiltrate*, fibrosis of muscularis propria*, noncaseating granuloma*.

* CD

Individuals with IBD should be classified into one of three categories, based on most recent diagnosis:

Crohn's disease (CD):

1. Evidence of small intestinal inflammation with endoscopically, radiologically or histologically demonstrated ulcerations, fistulation, mucosal fissuring, nodularity or cobblestoning, stricture formation or histologically demonstrated transmural inflammation with or without granuloma formation.
2. Isolated esophageal, gastric or duodenal inflammation with the finding of noncaseating granuloma.
3. Colonic inflammation which is patchy (normal segments separating areas of inflammation, as described above) or associated with one or more of the following features: complete rectal sparing, multiple (>10) aphthoid ulcers, deep ulceration (into the muscularis propria), transmural inflammation, extensive fibrosis and wall thickening, fistulation, non-caseating granuloma. (N.B. See note below regarding patchiness of endoscopically observed inflammation in patients with partially treated ulcerative colitis.)
4. The presence of complex suppurative perianal disease (i.e. more than a superficial fistula or uncomplicated superficial abscess).
5. If there are fewer than 10 aphthoid ulcers in the cecum (and the rest of the colon appears normal) in a patient with small bowel disease then this should be called small bowel disease only. Similarly, if the colon is normal except for the presence of a fistula extending from inflamed small bowel, the patient should be said to have small bowel disease alone. If the cecum is involved with ulcers larger than aphthoid ulcers or ulcers that are deep or if the involvement has resulted in deformity of the cecum this would be considered to be colonic involvement.

Ulcerative Colitis (UC)

1) Superficial inflammation and/or ulceration (involving only the mucosa and submucosa) of the colon which is continuous from the rectum extending proximally without skip lesions or complete rectal sparing (N.B. Relative rectal sparing is allowed for patients receiving topical rectal therapy; patchiness of endoscopic inflammation may be observed in patients with partially treated ulcerative colitis).

2) In patients with proctitis or left-sided ulcerative colitis there may be an area of inflammation in the cecum, usually surrounding the appendiceal orifice.

3) No inflammation of the small intestine ("backwash ileitis" is allowed - non-stricturing superficial inflammation of the terminal ileal mucosa associated with severe pancolitis which resolves following medical or surgical treatment of the colitis).

4) No features of Crohn's disease listed above.

Inflammatory Bowel Disease Unclassified (IBDU):

1. Confirmed IBD by A, B and C above.
2. Physician unable to classify individual into either CD or UC based on above criteria and/or patient has features of both CD and UC with none of the feature's diagnostic of one or the other.

Exclusion Criteria:

* 1.

Patients will be excluded if they meet any of the following criteria:

1. Inability to provide informed consent.
2. Non-English speaking
3. Patients presenting for a one-time consultation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with UC, CD, or IBDU starting Zymfentra (Infliximab-dyyb) in the setting of standard-of-care
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-11-20 (Actual); Primary Completion 2028-11-03 (Estimated); Study Completion 2028-11-03 (Estimated)

PRIMARY OUTCOMES:
Clinical remission as evaluated by the Simple Clinical Colitis Activity Index (SCCAI) for the patient-reported outcomes. | Weeks 0,1, 2, 4, 6,10, 14, 18, 24, 36, and 52.
  The SCCAI is a 6-item that describes the symptoms and disease activity of a patient with UC at the time of assessment. A score of 0-4 is considered a clinical range of remission (but with more refined definitions of clinical remission with SCCAI ≤2 and very mild symptoms with a score >2 ≤4), 5-7 mild activity, 8-16 moderate activity and > 16 severe activity. A response will be defined as a decrease of the SCCAI score < 5 points in patients with a baseline SCCAI ≥5.
Clinical remission as evaluated by the Simple Crohn's Disease Activity Index (sCDAI for the patient-reported outcomes. | Weeks 0,1, 2, 4, 6,10, 14, 18, 24, 36, and 52
  The Short Crohn's Disease Activity Index (sCDAI) is a simplified version of the Crohn's Disease Activity Index (CDAI), used to assess disease severity in Crohn's disease patients. It reduces the number of variables required, making it easier and quicker to use in clinical practice. Recent data demonstrated, that collections of the parameters on a single day equally reflects reliable disease activity compared to a collection of data over 7 consecutive days, which is often hampered by missing data.
  A score of < 150, 150-219, 220-450 and >450 reflects remission, mild, moderate and severe Crohn's disease activity.

SECONDARY OUTCOMES:
Response as measured by the Simple Endoscopic Score for Crohn's disease (SES-CD) | Through study completion, an average of 1 year
  The Simple Endoscopic Score for Crohn's Disease (SES-CD) is a tool used to objectively measure the severity of Crohn's disease based on the extent and severity of ulcers, affected surface area, and luminal narrowing during an endoscopy. The total score is the sum of scores for these four features, and it is categorized as follows: 0-2 for remission, 3-6 for mild activity, 7-15 for moderate activity, and greater than 15 for severe activity. Mucosal healing will be defined by an SES-CD < 4
Response as measured by the endoscopic Mayo score for ulcerative colitis | Through study completion, an average of 1 year
  The Mayo endoscopic score is a four-point scale (1 to 3) used to assess the severity of ulcerative colitis (UC) based on a colonoscopy. It evaluates the severity of inflammation through findings like erythema, vascular pattern, friability, erosions, and spontaneous bleeding, with higher scores indicating more severe disease. Mucosal healing will be defined by an endoscopic Mayo score <1.
Mucosal healing will be assessed in the setting of standard-of-care calprotectin levels. | Weeks 0, 14, 24, and 52.
  Calprotectin is a surrogate marker of intestinal inflammation, and levels ≥ 250 mcg/g stool are associated with active mucosal inflammation, whereas levels <150 mcg are considered to represent mild or no mucosal inflammation
Response as measured by Patient-Reported Outcomes Measurement Information System (PROMIS)- Depression | Weeks 0, 24, and 52.
  PROMIS measure of depression measures well-being. This is calculated as T scores. A clinically meaningful difference is considered to be a change in T score of ≥ 2.5 (scores are normalized at 50 with a standard deviation of 10). Higher scores mean more severe depression. Differences in PROMIS scores compared to baseline will be assessed.
Response as measured by Patient-Reported Outcomes Measurement Information System (PROMIS) -Anxiety Score | Weeks 0, 24, and 52.
  PROMIS measure of anxiety measures well-being. This is calculated as T scores. A clinically meaningful difference is considered to be a change in T score of ≥ 2.5 (scores are normalized at 50 with a standard deviation of 10). Higher scores indicate greater anxiety severity Differences in PROMIS scores compared to baseline will be assessed.
Response as measured by Patient-Reported Outcomes Measurement Information System (PROMIS) -Social Satisfaction Score | Weeks 0, 24, and 52.
  PROMIS measure of satisfaction measures well-being. This is calculated as T scores. A clinically meaningful difference is considered to be a change in T score of ≥ 2.5 (scores are normalized at 50 with a standard deviation of 10). Higher scores indicate greater satisfaction. Differences in PROMIS scores compared to baseline will be assessed.
Response as measured by Likert scale urgency Score | Weeks 0,1, 2, 4, 6,10, 14, 18, 24, 36, and 52
  Urgency will be measured by the 11-point Likert scale urgency question. Score range is 0-10. The higher the score, the worse the urgency.
Response as measured by Functional Assessment of Chronic Illness Therapy (FACIT)- Fatigue Scale Score | Weeks 0, 24, and 52
  Fatigue will be determined by the validated FACIT-F questionnaire. The FACIT-F is a 13-item measure that assesses self-reported fatigue and its impact upon daily activities and function. Score range is 0-52. The higher the score, the better the quality of life.
Response as measured by The Short Inflammatory Bowel Disease Questionnaire (SIBDQ) score | Weeks 0,4,10,14,18,24,36 and 52.
  The SIBDQ is a disease-specific health-related quality of life (HRQOL) questionnaire, able to detect and define meaningful clinical changes in inflammatory bowel disease (IBD) participants by measuring physical, social and emotional status. The SIBDQ consists of 10 questions; each question is scored on a scale from 1 (poor QOL) to 7 (optimum QOL). A higher score indicates a better health-related quality of life. Total scores range from 10 (poor QoL) to 70 (good QoL).
Response as measured by The Work Productivity and Activity Impairment questionnaire (WPAI) | Weeks 0, 24, and 52
  The WPAI was designed to measure absenteeism, presenteeism and activity impairment attributable to ill-health over the preceding 7 days. The WPAI calculates percentage impairment (maximum 100%) with higher numbers representing greater work impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Hans Herfarth, MD, PhD, Principal Investigator — University of North Carolina
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 3 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with the University of North Carolina [UNC].
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 36 months following article publication
Access Criteria: Researchers who provide a methodologically sound proposal.

REFERENCES:
- [Background] Popmihajlov Z, Pang L, Brown E, Joshi A, Su SC, Kaplan SS, Willis ED. A post hoc analysis utilizing the FDA toxicity grading scale to assess injection site adverse events following immunization with the live attenuated Zoster Vaccine (ZVL). Hum Vaccin Immunother. 2018;14(12):2916-2920. doi: 10.1080/21645515.2018.1502517. Epub 2018 Sep 5. PMID 30024827
- [Background] Youssef M, Hossein-Javaheri N, Hoxha T, Mallouk C, Tandon P. Work Productivity Impairment in Persons with Inflammatory Bowel Diseases: A Systematic Review and Meta-analysis. J Crohns Colitis. 2024 Sep 3;18(9):1486-1504. doi: 10.1093/ecco-jcc/jjae057. PMID 38647194
- [Background] Dubinsky MC, Panaccione R, Lewis JD, Sands BE, Hibi T, Lee SD, Naegeli AN, Shan M, Green LA, Morris N, Arora V, Bleakman AP, Belin R, Travis S. Impact of Bowel Urgency on Quality of Life and Clinical Outcomes in Patients With Ulcerative Colitis. Crohns Colitis 360. 2022 Jun 3;4(3):otac016. doi: 10.1093/crocol/otac016. eCollection 2022 Jul. PMID 36777426
- [Background] Singh S, Ananthakrishnan AN, Nguyen NH, Cohen BL, Velayos FS, Weiss JM, Sultan S, Siddique SM, Adler J, Chachu KA; AGA Clinical Guidelines Committee. Electronic address: clinicalpractice@gastro.org. AGA Clinical Practice Guideline on the Role of Biomarkers for the Management of Ulcerative Colitis. Gastroenterology. 2023 Mar;164(3):344-372. doi: 10.1053/j.gastro.2022.12.007. PMID 36822736
- [Background] Higgins PD, Schwartz M, Mapili J, Krokos I, Leung J, Zimmermann EM. Patient defined dichotomous end points for remission and clinical improvement in ulcerative colitis. Gut. 2005 Jun;54(6):782-8. doi: 10.1136/gut.2004.056358. PMID 15888785
- [Background] Peyrin-Biroulet L, Panes J, Sandborn WJ, Vermeire S, Danese S, Feagan BG, Colombel JF, Hanauer SB, Rycroft B. Defining Disease Severity in Inflammatory Bowel Diseases: Current and Future Directions. Clin Gastroenterol Hepatol. 2016 Mar;14(3):348-354.e17. doi: 10.1016/j.cgh.2015.06.001. Epub 2015 Jun 11. PMID 26071941
- [Background] Thia K, Faubion WA Jr, Loftus EV Jr, Persson T, Persson A, Sandborn WJ. Short CDAI: development and validation of a shortened and simplified Crohn's disease activity index. Inflamm Bowel Dis. 2011 Jan;17(1):105-11. doi: 10.1002/ibd.21400. PMID 20629100
- [Background] Barnes EL, Hanson JS, Regueiro MD, Saha S, Sands BE, Rubin DT, Dubinsky MC, Siegel CA, Gazis DR, Crawford JM, Long MD. Older Adult Patients Use More Aminosalicylate Monotherapy Compared With Younger Patients With Inflammatory Bowel Disease: TARGET-IBD. J Clin Gastroenterol. 2022 Jul 1;56(6):529-535. doi: 10.1097/MCG.0000000000001557. Epub 2021 Jun 11. PMID 34115661
- [Background] Reilly MC, Zbrozek AS, Dukes EM. The validity and reproducibility of a work productivity and activity impairment instrument. Pharmacoeconomics. 1993 Nov;4(5):353-65. doi: 10.2165/00019053-199304050-00006. PMID 10146874
- [Background] Tinsley A, Macklin EA, Korzenik JR, Sands BE. Validation of the functional assessment of chronic illness therapy-fatigue (FACIT-F) in patients with inflammatory bowel disease. Aliment Pharmacol Ther. 2011 Dec;34(11-12):1328-36. doi: 10.1111/j.1365-2036.2011.04871.x. Epub 2011 Oct 17. PMID 21999576
- [Background] Adegbola SO, Dibley L, Sahnan K, Wade T, Verjee A, Sawyer R, Mannick S, McCluskey D, Bassett P, Yassin N, Warusavitarne J, Faiz O, Phillips R, Tozer PJ, Norton C, Hart AL. Development and initial psychometric validation of a patient-reported outcome measure for Crohn's perianal fistula: the Crohn's Anal Fistula Quality of Life (CAF-QoL) scale. Gut. 2021 Sep;70(9):1649-1656. doi: 10.1136/gutjnl-2019-320553. Epub 2020 Dec 3. PMID 33272978
- [Background] Dubinsky MC, Clemow DB, Hunter Gibble T, Li X, Vermeire S, Hisamatsu T, Travis SPL. Clinical Effect of Mirikizumab Treatment on Bowel Urgency in Patients with Moderately to Severely Active Ulcerative Colitis and the Clinical Relevance of Bowel Urgency Improvement for Disease Remission. Crohns Colitis 360. 2022 Dec 13;5(1):otac044. doi: 10.1093/crocol/otac044. eCollection 2023 Jan. PMID 36777368
- [Background] Long MD, Afzali A, Fischer M, Hudesman D, Abdalla M, McCabe R, Cohen BL, Ungaro RC, Harlan W, Hanson J, Konijeti G, Polyak S, Ritter T, Salzberg B, Seminerio J, English E, Zhang X, Sharma PP, Herfarth HH. Tofacitinib Response in Ulcerative Colitis (TOUR): Early Response After Initiation of Tofacitinib Therapy in a Real-world Setting. Inflamm Bowel Dis. 2023 Apr 3;29(4):570-578. doi: 10.1093/ibd/izac121. PMID 35700276
- [Background] Irvine EJ, Zhou Q, Thompson AK. The Short Inflammatory Bowel Disease Questionnaire: a quality of life instrument for community physicians managing inflammatory bowel disease. CCRPT Investigators. Canadian Crohn's Relapse Prevention Trial. Am J Gastroenterol. 1996 Aug;91(8):1571-8. PMID 8759664
- [Background] Bewtra M, Brensinger CM, Tomov VT, Hoang TB, Sokach CE, Siegel CA, Lewis JD. An optimized patient-reported ulcerative colitis disease activity measure derived from the Mayo score and the simple clinical colitis activity index. Inflamm Bowel Dis. 2014 Jun;20(6):1070-8. doi: 10.1097/MIB.0000000000000053. PMID 24810138
- [Background] Henao MP, Bewtra M, Osterman MT, Aberra FN, Scott FI, Lichtenstein GR, Kraschnewski J, Lewis JD. Measurement of Inflammatory Bowel Disease Symptoms: Reliability of an Abbreviated Approach to Data Collection. Inflamm Bowel Dis. 2015 Oct;21(10):2262-71. doi: 10.1097/MIB.0000000000000496. PMID 26193348
- [Background] Satsangi J, Silverberg MS, Vermeire S, Colombel JF. The Montreal classification of inflammatory bowel disease: controversies, consensus, and implications. Gut. 2006 Jun;55(6):749-53. doi: 10.1136/gut.2005.082909. PMID 16698746
- [Background] Hanauer SB, Sands BE, Schreiber S, Danese S, Klopocka M, Kierkus J, Kulynych R, Gonciarz M, Soltysiak A, Smolinski P, Sreckovic S, Valuyskikh E, Lahat A, Horynski M, Gasbarrini A, Osipenko M, Borzan V, Kowalski M, Saenko D, Sardinov R, Lee SJ, Kim S, Bae Y, Lee S, Lee S, Lee JH, Yang S, Lee J, Lee J, Kim JM, Park G, Sandborn WJ, Colombel JF. Subcutaneous Infliximab (CT-P13 SC) as Maintenance Therapy for Inflammatory Bowel Disease: Two Randomized Phase 3 Trials (LIBERTY). Gastroenterology. 2024 Oct;167(5):919-933. doi: 10.1053/j.gastro.2024.05.006. Epub 2024 May 23. PMID 38788861
- [Background] Church PC, Hyams J, Ruemmele F, de Ridder L, Turner D, Griffiths AM. The Continental Divide: Anti-TNF Use in Pediatric IBD Is Different in North America Compared to Other Parts of the World. Can J Gastroenterol Hepatol. 2018 Jun 12;2018:3190548. doi: 10.1155/2018/3190548. eCollection 2018. PMID 30009157
- [Background] Horst SN, Kirkpatrick M, Scoville E, Buisson A. How to Incorporate Subcutaneous Infliximab and Vedolizumab in Your Practice. Clin Gastroenterol Hepatol. 2025 Feb;23(2):216-219.e2. doi: 10.1016/j.cgh.2024.07.042. Epub 2024 Oct 8. No abstract available. PMID 39393781
- [Background] Roblin X, Veyrard P, Bastide L, Berger AE, Barrau M, Paucelle AS, Waeckel L, Kwiatek S, Flourie B, Nancey S, Paul S. Subcutaneous injection of infliximab CT-P13 results in stable drug levels within 14-day treatment cycle in Crohn's disease. Aliment Pharmacol Ther. 2022 Jul;56(1):77-83. doi: 10.1111/apt.16852. Epub 2022 Feb 28. PMID 35229331
- [Background] Roblin X, Nancey S, Papamichael K, Duru G, Flamand M, Kwiatek S, Cheifetz A, Fabien N, Barrau M, Paul S. Higher Serum Infliximab Concentrations Following Subcutaneous Dosing are Associated with Deep Remission in Patients with Inflammatory Bowel Disease. J Crohns Colitis. 2024 May 31;18(5):679-685. doi: 10.1093/ecco-jcc/jjad188. PMID 37934041
- [Background] Iborra M, Caballol B, Garrido A, Huguet JM, Mesonero F, Ponferrada A, Arias Garcia L, Bosca Watts MM, Fernandez Prada SJ, Brunet Mas E, Gutierrez Casbas A, Cerrillo E, Ordas I, Ruiz L, Garcia de la Filia I, Escobar Ortiz J, Sicilia B, Ricart E, Domenech E, Nos P. Subcutaneous Infliximab Cutoff Points in Patients With Inflammatory Bowel Disease: Data From the ENEIDA Registry. J Crohns Colitis. 2025 Jan 11;19(1):jjae127. doi: 10.1093/ecco-jcc/jjae127. PMID 39171615
- [Background] Outtier A, Gijbels L, Noman M, Verstockt B, Sabino J, Vermeire S, Ferrante M. Screening Failure in a Large Clinical Trial Centre for Inflammatory Bowel Diseases: Rates, Causes, and Outcomes. Inflamm Bowel Dis. 2023 Sep 1;29(9):1440-1445. doi: 10.1093/ibd/izac227. PMID 36350998
- [Background] Ha C, Ullman TA, Siegel CA, Kornbluth A. Patients enrolled in randomized controlled trials do not represent the inflammatory bowel disease patient population. Clin Gastroenterol Hepatol. 2012 Sep;10(9):1002-7; quiz e78. doi: 10.1016/j.cgh.2012.02.004. Epub 2012 Feb 15. PMID 22343692
- [Background] Dulai PS, Singh S, Jairath V, Wong E, Narula N. Integrating Evidence to Guide Use of Biologics and Small Molecules for Inflammatory Bowel Diseases. Gastroenterology. 2024 Mar;166(3):396-408.e2. doi: 10.1053/j.gastro.2023.10.033. Epub 2023 Nov 8. PMID 37949249
- [Background] Lichtenstein GR, Yan S, Bala M, Hanauer S. Remission in patients with Crohn's disease is associated with improvement in employment and quality of life and a decrease in hospitalizations and surgeries. Am J Gastroenterol. 2004 Jan;99(1):91-6. doi: 10.1046/j.1572-0241.2003.04010.x. PMID 14687148
- [Background] Ananthakrishnan AN, Weber LR, Knox JF, Skaros S, Emmons J, Lundeen S, Issa M, Otterson MF, Binion DG. Permanent work disability in Crohn's disease. Am J Gastroenterol. 2008 Jan;103(1):154-61. doi: 10.1111/j.1572-0241.2007.01561.x. Epub 2007 Dec 11. PMID 18076736
- [Background] Shivashankar R, Tremaine WJ, Harmsen WS, Loftus EV Jr. Incidence and Prevalence of Crohn's Disease and Ulcerative Colitis in Olmsted County, Minnesota From 1970 Through 2010. Clin Gastroenterol Hepatol. 2017 Jun;15(6):857-863. doi: 10.1016/j.cgh.2016.10.039. Epub 2016 Nov 14. PMID 27856364
- [Background] Herrinton LJ, Liu L, Lewis JD, Griffin PM, Allison J. Incidence and prevalence of inflammatory bowel disease in a Northern California managed care organization, 1996-2002. Am J Gastroenterol. 2008 Aug;103(8):1998-2006. doi: 10.1111/j.1572-0241.2008.01960.x. PMID 18796097
- [Background] Loftus EV Jr, Schoenfeld P, Sandborn WJ. The epidemiology and natural history of Crohn's disease in population-based patient cohorts from North America: a systematic review. Aliment Pharmacol Ther. 2002 Jan;16(1):51-60. doi: 10.1046/j.1365-2036.2002.01140.x. PMID 11856078